CLINICAL TRIAL: NCT03747406
Title: Comparison Between Ultrasound-guided Erector Spinae Block and Transverse Abdominis Plane Block in Obese Patients Undergoing Sleeve Gasterectomy.
Brief Title: Erector Spinae Block and Transverse Abdominis Plane Block for Sleeve Gasterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dalia Ismail (Other)
Collaborators: Abdelhamid, Bassant Mohamed, M.D. (Individual)
Responsible Party: Sponsor-Investigator, Dalia Ismail, Lecturer of Anaesthesia- Cairo University, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: N-125-2018
Record Dates: First submitted 2018-11-14; First posted 2018-11-20 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Bariatric Surgery Candidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ESP group (Experimental): The patient rolled to his side, the level between T9 and T10 identified using ultrasound. An 8-14 MHz curved array probe (Siemens ACUSON X300 Ultrasound System) will be applied longitudinal orientation 3 cm lateral midline. The erector spinae and the psoas muscle will be identified. A skin wheal will be made using lidocaine 1% at each level and then a 22-gauge, 8 cm Tuohy needle (Perifix Epidural Needle) will be advanced inplane until contact with the transverse process. The needle will be withdrawn slightly and 30cc of bupivacaine 0.25 % (15ml for each side) will be injected slowly after negative aspiration confirmed. The same procedure will be repeated in the contralateral side.
  Interventions: Procedure: Erector spinae plane block
- TAP group (Experimental): The patient in supine position. Under complete aseptic conditions, a linear array transducer 5-12 MHz (Siemens ACUSON X300 Ultrasound System) will be positioned inferior and parallel to the costal margin in a medio-lateral orientation. The external oblique, internal oblique and transverse abdominis muscles will be identified immediately lateral to the linea semilunaris. A a 22-gauge, 8 cm Tuohy needle (Perifix Epidural Needle) will be advanced medially and in-plane to the US beam until the tip lies between the fascia of the internal oblique muscle and the transverse abdominis muscle layers. 30 ml of 0.25 % bupivacaine will be injected in each side and the spread will be observed between the two muscles layers.
  Interventions: Procedure: TAP block
- opioid group (No Intervention): will receive intravenous morphine with general anesthesia and total opioid consumption will be calculated

INTERVENTIONS:
Procedure: Erector spinae plane block — the level between T9 and T10 will be identified using ultrasound as well as transverse processes depth. An array probe will be applied longitudinal orientation 3 cm lateral midline. The erector spinae and the psoas muscle will be identified. A skin wheal will be made using lidocaine 1% at each level and then a 22-gauge Tuohy needle will be advanced inplane until it made contact with the transverse process. The needle will be withdrawn slightly and 30cc of bupivacaine 0.25 % (15ml for each side) will be injected slowly after negative aspiration was confirmed. The same procedure will be repeated in the contralateral side.
  Arms: ESP group
Procedure: TAP block — a linear array transducer 5-12 MHz will be positioned inferior and parallel to the costal margin in a medio-lateral orientation. The external oblique, internal oblique and transverse abdominis muscles will be identified immediately lateral to the linea semilunaris. A a 22-gauge needle will be advanced medially and in-plane to the US beam until the tip lies between the fascia of the internal oblique muscle and the transverse abdominis muscle layers. 30 ml of 0.25 % bupivacaine will be injected in each side and the spread will be observed between the two muscles layers.
  Arms: TAP group

SUMMARY:
assess the efficacy of ultrasound guided erector spinae block to decrease the requirement for analgesics after laparoscopic sleeve gastrectomy and to decrease postoperative pain scores and opioid consumption compared to subcostal transverses abdominis block.

DETAILED DESCRIPTION:
Primary outcomes

• Cumulative opioid consumption during the first 24 h postoperatively. For the purpose of comparison, all opioids administered postoperatively will be converted to IV morphine equivalent doses using standard opioid dosage conversion tables.

Secondary outcome parameters

1. Pain assessment by the aid of Visual analogue scale (VAS), which is consisted of a "10 cm" line with one end labeled no pain and other end labeled worst intolerable pain. The patients marked the line at the point that best describing the pain intensity. The preoperative assessment included training of the patients about (VAS) for postoperative pain. The length of the line to the patient's mark will be measured and recorded postoperative after 30 min., 4, 6, 8, and 24 hours.
2. Failure rate of the block will be calculated, where the block will be considered a failed block if the patient requires more than two doses of rescue analgesia in the first hour postoperatively.
3. Duration of surgery (from skin incision till skin closure) and general anesthesia (from induction of GA till extubation).
4. Incidence of complications, such as: Nerve injury, Hematoma formation, LA toxicity, and intravascular injection.

ELIGIBILITY:
Inclusion Criteria:

* • Patients from 18 to 59 years.

  * BMI > 40 kg/m2
  * Genders eligible for study: both.
  * ASA I-III.
  * No contraindications for application of regional anesthesia as Patient refusal, local anesthetic allergy, local sepsis or infection at puncture site, INR > 1.5 or < 12 hours post LMWH.

Exclusion Criteria:

* • Patient refusal.

  * Extremes of age.
  * ASA IV.
  * Increased intracranial pressure.
  * Coagulopathy or thrombocytopenia less than 100000/ml.
  * Sepsis (increased risk of meningitis).
  * Infection at the puncture site.
  * Pre-existing neurologic disease.
  * History of allergy to local anesthetic.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
Cumulative opioid consumption during the first 24 h postoperatively | 24 hours after surgery
  measure total opioid dose in 24 hours after surgery

SECONDARY OUTCOMES:
pain assessment by Visual Analog Scale | 24 hours after surgery
  it is a "10 cm" line with one end labeled no pain and other end labeled worst intolerable pain. The patients marked the line at the point that best describing the pain intensity. The preoperative assessment included training of the patients about (VAS) for postoperative pain. The length of the line to the patient's mark will be measured and recorded postoperative after 30 min., 4, 6, 8, and 24 hours.If the VAS level is 5 or more this means failure of analgesio and a dose of rescue analgesia is given

CONTACTS AND LOCATIONS:
Overall Officials: Bassant M Abdelhamid, MD, Principal Investigator — Cairo University; Dalia Khaled, MD, Study Director — Cairo University
Locations (1):
- Faculty of Medicine - Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No